CLINICAL TRIAL: NCT07355283
Title: A Randomized, Double-Blind, Controlled, Multicenter, Phase III Clinical Study of IMM0306 (Amulirafusp Alfa) for Injection in Combination With Lenalidomide Versus Placebo in Combination With Lenalidomide in Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: IMM0306 in Combination With Lenalidomide vs Placebo in Combination With Lenalidomide in Patients With Relapsed/Refractory Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMM0306-004
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMM0306 in combination with lenalidomide (Experimental): One treatment cycle consists of 4 weeks (28 days). IMM0306 (Amulirafusp Alfa) will be administered once weekly, and lenalidomide will be administered from Day 1 to Day 21 of each cycle.
  Interventions: Drug: IMM0306 2.0 mg/kg; Drug: Lenalidomide 20 mg
- Placebo in combination with lenalidomide (Placebo Comparator): One treatment cycle consists of 4 weeks (28 days). Placebo will be administered once weekly, and lenalidomide will be administered from Day 1 to Day 21 of each cycle.
  Interventions: Drug: Placebo; Drug: Lenalidomide 20 mg

INTERVENTIONS:
Drug: IMM0306 2.0 mg/kg — IV infusion;
  Other Names: Amulirafusp Alfa
  Arms: IMM0306 in combination with lenalidomide
Drug: Placebo — IV infusion;
  Arms: Placebo in combination with lenalidomide
Drug: Lenalidomide 20 mg — orally

SUMMARY:
This study is a randomized, controlled, double-blind, multicenter, phase III clinical study to evaluate the efficacy of IMM0306 (Amulirafusp Alfa)in combination with lenalidomide versus placebo in combination with lenalidomide in patients with Relapsed/Refractory Follicular lymphoma. Primary endpoints are Complete Remission Rate (CRR) and Progression-Free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
2. At least one measurable lesion (as per Lugano 2014 criteria).
3. Histologically confirmed CD20-positive Follicular Lymphoma, Grade 1, 2, or 3a.
4. Previously received at least two prior systemic regimens, including at least one line containing an anti-CD20 monoclonal antibody.
5. Adequate hepatic, hematologic, and renal function.
6. Expected survival at least 6 months.

Exclusion Criteria:

1. Autologous HSCT within 100 days prior to first administration, or any prior allogeneic HSCT or solid organ transplantation.
2. History of central nervous system (CNS) metastases or active CNS involvement.
3. History of other malignancy within the past 5 years.
4. Severe organic cardiovascular or cerebrovascular diseases.
5. History of severe allergic reactions to any components of the trial drug, any macromolecular protein preparations or monoclonal antibodies.
6. Previous treatment with anti-CD47 monoclonal antibody/SIRPα fusion protein.
7. Human immunodeficiency virus (HIV) infection.
8. Echocardiography examination indicating left ventricular ejection fraction (LVEF) < 55%.
9. Active infection requiring systemic therapy (e.g., fungal, bacterial, viral).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate(CRR) as Assessed by Investigator | approximately 48 months
  CRR is defined as the percentage of participants who achieve a CR(Complete Response) determined per Lugano 2014 criteria (2014 Lugano Revised Response Criteria for Malignant Lymphoma).
Progression-Free Survival (PFS) as Assessed by Investigator | approximately 48 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Complete remission rate(CRR) as Assessed by Independent Review Committee(IRC) | approximately 48 months
  CRR is defined as the percentage of participants who achieve a CR determined per Lugano 2014 criteria.
Progression-Free Survival (PFS) as Assessed by Independent Review Committee(IRC) | approximately 48 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | approximately 48 months
  ORR is defined as the proportion of the analysis population achieving CR, PR(Partial Response).
Duration of Response (DOR) | approximately 48 months
  DOR is defined as the time from the first documented evidence of complete response or partial response until disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | approximately 60 months
  OS is defined as the time from randomization to death due to any cause.
Time to Next Anti-Lymphoma Treatment(TTNT) | approximately 48 months
  TTNT is defined as the number of days from randomization to the date of next anti-lymphoma treatment.
Adverse Event (AE) | approximately 48 months
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No